CLINICAL TRIAL: NCT04794387
Title: The Lymphoma and Leukemia Society Amended COVID-19 Registry
Status: Completed | Type: Observational
Sponsor: Blood Cancer United (Other)
Responsible Party: Sponsor
Other Study IDs: LLSC19-001-Amendment 1
Record Dates: First submitted 2021-03-09; First posted 2021-03-12 (Actual); Last update posted 2023-03-02 (Actual); Status verified 2021-08

CONDITIONS: Covid19
Keywords: COVID-19 Booster
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Biological: Amended LLS COVID-19 Registry — Do people with blood cancer who did not develop antibodies after a complete COVID-19 vaccination, develop antoibodies after a COVID-19 booster?

SUMMARY:
The LLS COVID-19 Registry is being amended to invite people who participated in the LLS COVID-19 Registry and did not develop antibodies after receiving a complete COVID-19 vaccination, as well as people with blood cancer who did not participate in the initial LLS COVID-19 Registry and also did not develop antibodies after receiving a complete COVID-19 vaccination, to participate in this amended LLS COVID-19 Registry.

DETAILED DESCRIPTION:
The results of the Leukemia and Lymphoma Society (LLS) COVID-19 Registry indicate that about twenty-five percent (25%) of people with blood cancer and on immunosuppressants participating in the LLS COVID-19 Registry, who received a complete COVID-19 vaccination, did not develop antibodies.

The Food and Drug Administration has authorized third doses (boosters) of the Pfizer and Moderna Covid-19 vaccines for people with weakened immune systems, in a bid to bolster their protection against infection as the highly contagious Delta variant circulates. The agency will amend the emergency-use authorizations for the two vaccines to allow immunocompromised people to get an additional dose.

Therefore the LLS COVID-19 Registry is being amended to invite people who participated in the LLS COVID-19 Registry and did not develop antibodies as noted above, as well as people with blood cancer who did not participate in the initial LLS COVID-19 Registry and also did not develop antibodies after receiving a complete COVID-19 vaccination, to participate in this amended LLS COVID-19 Registry. Using the same design as the initial COVID-19 Registry (Protocol LLSC19-001), this amended LLS COVID-19 Registry will determine if people who have decided to receive a booster vaccination, who did not develop antibodies after receiving a complete COVID-19 vaccination will develop antibodies after a single dose booster of either the Pfizer or Moderna COVID-19 vaccination.

ELIGIBILITY:
Inclusion Criteria:

* People with blood cancer who did not develop antibodies after a complete COVID-19 vaccination.

Exclusion Criteria:

* People who receiived a complete COVID-19 vaccination and did develop antibodies.
* People unwilling or unable to receive COVID-19 booster.

Min Age: 21 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: People with blood cancer who did not develop antibodies after a complete COVID-19 vaccination.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2021-08-27 (Actual); Primary Completion 2022-12-13 (Actual); Study Completion 2022-12-13 (Actual)

PRIMARY OUTCOMES:
A SARS antibody test will be paired with surveys to measure the response people with blood cancer, who did not develop antibodes after a complete COVID-19 vaccination, have to the COVID-19 booster. | 10 years
  Observational Study

CONTACTS AND LOCATIONS:
Locations (1):
- Lymphoma and Leukemia Society, Rye Brook, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
ONLY De-identified data will be made available to researchers approved by The Lymphoma and Leukemia Society.
Supporting Information: Study Protocol
Time Frame: data will become available after it is de-identified and entered into a secure database. This data will be collected and made available over 10 years.